CLINICAL TRIAL: NCT04009083
Title: CLINICAL UTILITY OF AXUMIN PET/MRI IMAGING TWO YEARS FOLLOWING FOCAL CRYO-ABLATION (FCA) OF PROSTATE CANCER
Brief Title: Axumin PETMRI Imaging Following Focal Cryo-ablation (FCA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-00123
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer
Keywords: 18F-Fluciclovine PET imaging; Focal Cryo Ablation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Other)
  Interventions: Device: Standard of Care MRI
- 18F-Fluciclovine PET Scan (Experimental)
  Interventions: Other: Fluciclovine PET scan added to MRI

INTERVENTIONS:
Device: Standard of Care MRI — Prostate MRI, serum Prostate Specific Antigen (PSA), in field and random systemic prostate biopsies
  Arms: Standard of Care
Other: Fluciclovine PET scan added to MRI — 18F-Fluciclovine (Axumin) is a radioactive diagnostic agent indicated for positron emission tomography (PET) imaging in men with suspected prostate cancer recurrence based on elevated blood prostate specific antigen (PSA) levels following prior treatment
  Arms: 18F-Fluciclovine PET Scan

SUMMARY:
This is a prospective outcomes study assessing quality of life and oncological control at pre-defined time points following FOCAL CRYO-ABLATION (FCA). The investigator's standard of care is to perform an Magentic Resonance Imaging (MRI) and prostate biopsy two years following FCA. The prostate biopsy assesses both the presence of in field and out of field disease. The role of Axumin PET/MRI for detecting disease following FCA has not been previously examined.

DETAILED DESCRIPTION:
The primary hypothesis of this study is that 18F-Fluciclovine PET/MRI imaging at two years following FCA will improve sensitivity for detection of in field recurrence of significant prostate cancer defined as any Gleason pattern 4 disease.

The secondary hypothesis of this study is that 18F-Fluciclovine PET/MRI imaging at two years following FCA will improve sensitivity for detection of out of field recurrence of significant prostate cancer .

ELIGIBILITY:
Inclusion Criteria:

* FCA at NYU Langone Health performed at least two years prior to study enrollment by Drs. Lepor or Wysock.
* No prostate cancer specific treatment following FCA
* Consented to undergo reflex MRI and prostate biopsy two years following FCA.

Exclusion Criteria:

* Any contraindication to prostate biopsy
* Prior allergic reaction to 18F-Fluciclovine
* Patient refuses MRI and prostate biopsy two years following FCA.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

PRIMARY OUTCOMES:
Measure of sensitivity following PET imaging with 18-F fluciclovine (Axumin) | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Lepor, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States